CLINICAL TRIAL: NCT04638725
Title: Identification of Genetic Determinants for Treatment Resistance/Sensitivity and/or Toxicity in Adjuvant Setting for HER2 Positive Breast Cancer
Acronym: SIGHER
Status: Recruiting | Type: Observational
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-010
Record Dates: First submitted 2020-11-09; First posted 2020-11-20 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — Blood Specimen Collection; Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood sample, Tumour paraffin-embedded sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- HER2 positive breast cancer treated only with trastuzumab
  Interventions: Other: Blood sample for genetic analysis
- HER2 positive breast cancer treated with pertuzumab
  Interventions: Other: Blood sample for genetic analysis
- HER2 positive breast cancer treated with neratinib
  Interventions: Other: Blood sample for genetic analysis
- HER2 positive breast cancer treated with Trastuzumab emtansine (TDM1)
  Interventions: Other: Blood sample for genetic analysis
- HER2 positive breast cancer treated with TDM1 and neratinib
  Interventions: Other: Blood sample for genetic analysis

INTERVENTIONS:
Other: Blood sample for genetic analysis — Blood samples will be collected in two 6 ml EDTA tubes after informed consent and inclusion in the study

SUMMARY:
This is a multicenter, non-randomized, prospective cohort study. The purpose of the study is to identify constitutional genetic factors associated with histological response, resistance or sensibility to treatment in human epidermal growth factor receptor 2 (HER2)-positive breast cancer. 9000 patients will be enrolled in this study. Blood samples will be collected after informed consent and inclusion in the study. Patients will be treated and followed according to the standards of their treating center. They will be followed every six months for five years.

DETAILED DESCRIPTION:
The purpose of the SIGHER trial is to create a cohort of 9000 patients with HER2-positive breast cancer including detailed epidemiologic and treatment data. The distribution of constitutional genetic variants will be evaluated within groups of patients treated with different regimes of targeted therapies, identifying variants associated with histological response, as well as sensitivity or resistance to these therapies.

Blood samples will be collected in two 6ml ethylenediaminetetraacetic acid (EDTA) tubes after informed consent and inclusion in the study.

As the samples are received at the biological resource center, total blood will be aliquoted into a 500 µl tube and frozen at -80° C. DNA will be extracted using standard protocols. DNA will be stored in anticipation of genetic analyses. An aliquot of the DNA sample will be genotyped for a panel of high-density genetic markers covering the whole genome for genome-wide association studies.

ELIGIBILITY:
For inclusion in the study, patients must be affiliated to the national or local social security, and must meet all the following criteria:

Inclusion Criteria:

* Age ≥ 18 years
* Histological diagnosis of breast adenocarcinoma. Non-metastatic and operable.
* Current or prior treatment with one therapy targeting HER2 in adjuvant or neoadjuvant phase for the current breast cancer
* Given written informed consent

Exclusion Criteria:

* Patients not able to comply to the protocol assessments for geographic, social or psychological reasons
* Patients placed under judicial protection, guardianship, or supervision
* History of cancer in the 5 years preceding anti-HER2 therapy initiation
* Concomitant cancer (except for an other non metastatic cancer treated only with surgery)

Note : Patients are eligible at any time of the follow-up if the adjuvant or neoadjuvant chemotherapy started after 01/01/2019. Patients treated with trastuzumab, pertuzumab, neratinib or T-DM1 in a clinical trial are eligible in the SIGHER study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2-positive Breast Cancer
Sampling Method: Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2029-12-15 (Estimated); Study Completion 2029-12-15 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) | at the end of enrollment (3 years)
  Constitutional genetic variants using a genome-wide approach will be tested for association with pCR as a function of neoadjuvant treatment targeting HER2.
Disease Free Survival (DFS) | At the end of the study (8 years)
  Constitutional genetic variants using a genome-wide approach will be tested for association with DFS as a function of treatment
Overall Survival (OS) | At the end of the study (8 years)
  Constitutional genetic variants using a genome-wide approach will be tested for association with OS as a function of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France